CLINICAL TRIAL: NCT02789930
Title: Evaluation of a Program for Length Based Weight Estimation in Comparison to the Anesthesia Tape ("Anästhesie-Lineal")
Brief Title: Evaluation of Program for Length Based Weight Estimation
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2015-0191 - Part 3
Record Dates: First submitted 2016-05-30; First posted 2016-06-03 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Length-based Weight Estimation; Body Weights and Measures
Keywords: Weight estimation; Patient safety
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Device: Accuracy of a program and the anesthesia tape ("Anästhesie-Lineal") — Computer based comparison of the two devices based on collected patient data

SUMMARY:
The purpose of this prospective single center study is to investigate if a developed program is more accurate than the anesthesia tape ("Anästhesie-Lineal"). For this study 1000 patients are required to collect anonymized data (length, weight, age, anesthesia material used during anesthesia) for achieving a power of 80% during statistical analysis. The main hypothesis ist that the program has a better accuracy than the anesthesia tape ("Anästhesie-Lineal").

DETAILED DESCRIPTION:
This prospective single center study is performed at the university children's Hospital zurich. Patients planned for surgery in general anesthesia with intubation, aged 0 to 16 years and with a body length suitable for the emergency tapes can be included in this study. Patient and parental information is performed during the pre-anesthetic visit. After written consent the patient will be included. Patient ́s length and weight will be measures earliest one day before data collection. Data collection during anesthesia has no influence on the daily anesthesia routine and has no impact on patient safety and anaesthesia. Patient's data is made anonymous for further inspection. Data is documented in Microsoft Excel and statistical analysis calculated with SPSS. 1000 patients are needed for a power of 80%. Primary outcome parameter is length based weight estimation, secondary outcome parameters are length based age estimation and the correctness of recommended anesthesia material (endotracheal tube, laryngeal mask, oropharyngeal mask and face mask). Both tools (program and anesthesia tape ["Anästhesie-Lineal"]) will be compared with each other regarding primary and secondary outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* body length suitable with the investigated emergency tapes
* all patients aged 0 -16 years
* receiving general anesthesia with intubation or laryngeal mask

Exclusion Criteria:

* Already included in this study once
* missing patient or parental consent

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients planned for elecitve surgery in general anesthesia
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
length-based weight-estimation by program | intraoperative
  The by the program estimated bodyweight based on the patient's Body length is investigated regarding the estimations accuracy and cases in the +/- 10% interval

SECONDARY OUTCOMES:
length based age estimation | intraoperative
  The by the program estimated age based on the patient's body length is investigated regarding the estimations accuracy
size of endotracheal tube | intraoperative
  The by the program suggested endotracheal tube based on the patient's Body length is investigated regarding the correctness
size of laryngeal mask | intraoperative
  The by the program suggested laryngeal mask based on the patient's Body length is investigated regarding the correctness
size of facemask | intraoperative
  The by the program suggested facemask based on the patient's body length is investigated regarding the correctness
size of oropharyngeal tube | intraoperative
  The by the program suggested oropharyngeal tube based on the patient's Body length is investigated regarding the correctness

CONTACTS AND LOCATIONS:
Overall Officials: Achim J Schmitz, M.D., Study Chair — University Children's Hospital, Zurich
Locations (1):
- University Childrens Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided